CLINICAL TRIAL: NCT06870305
Title: Efficacy of Mindfulness in PREventing Progression to Psychosis in Individuals With an Ultra High Risk for Psychosis
Acronym: EM-PREPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Psychothérapique de Nancy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-A02766-39; RIPH 2023-04 (Other: centre Psychothérapique de Nancy CPN)
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Clinical High Risk for Psychosis (CHR)
Keywords: Psychosis; mindfulness
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MBTP group (Experimental)
  Interventions: Other: MBTP : Mindflulness based training for psychosis
- TAU group (No Intervention)

INTERVENTIONS:
Other: MBTP : Mindflulness based training for psychosis — The group-based mindfulness programme is called MBTP (Mindfulness based training for psychosis). The MBTP programme consists of 5 sessions over a period of one month (2 sessions in the first week, then one session a week). Each session lasts approximately 1h30 and is carried out in a group of 5 participants. The sessions cover informal and formal mindfulness tasks, elements of psycho-education on emotions, meditation exercises on emotions, and thought defusion and acceptance tasks. Participants are encouraged to meditate at home between sessions.
  Arms: MBTP group

SUMMARY:
The main objective is to evaluate the efficacy of a group-based mindfulness therapy programme in reducing distress associated with symptoms of UHR (Ultra High Risk) or FEP (first psychotic episode) compared with usual treatment. The secondary objectives were to study the efficacy of a group-based mindfulness intervention: on the reduction of psychotic symptoms; on the maintenance over time (6 months of follow-up) of the efficacy of the intervention on the distress associated with the symptoms of the UHR or PEP state; and on various dimensions associated with care: cognitive functions, anxiety, quality of life.

ELIGIBILITY:
Inclusion Criteria:

* People aged between 18 and 30 validating the criteria for UHR or PEP status on the CAARMS scale and having a social functional impact (SOFAS score below 50 or a reduction of more than 30% in the score)

Exclusion Criteria:

* Previous episode of schizophrenic disorder, schizoaffective disorder or bipolar disorder
* Previous antipsychotic treatment for more than 12 months
* Organic mental disorder or intellectual disability
* Serious suicidal/homicidal risk (but admissible if this risk has been resolved)
* Insufficient French language skills
* Adult incapable of giving consent and not under legal protection
* Protection measure (guardianship/curatorship/court supervision) or under court supervision
* Person deprived of liberty by judicial or administrative decision (including forced hospitalisation)
* Persons in a life-threatening emergency
* Not affiliated to a social security regime

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Distress related to psychotic symptoms | 3 months
  Distress related to psychotic symptoms on the CAARMS scale at the end of therapeutic intervention
Distress related to psychotic symptoms | 4 months
  Distress related to psychotic symptoms on the CAARMS scale at the end of therapeutic intervention
Distress related to psychotic symptoms | 6 months
  Distress related to psychotic symptoms on the CAARMS scale at the end of therapeutic intervention
Distress related to psychotic symptoms | 9 months
  Distress related to psychotic symptoms on the CAARMS scale at the end of therapeutic intervention

SECONDARY OUTCOMES:
Intensity of psychotic symptoms | 3 months
  Intensity of psychotic symptoms on the CAARMS scale
Intensity of psychotic symptoms | 4 months
  Intensity of psychotic symptoms on the CAARMS scale
Intensity of psychotic symptoms | 6 months
  Intensity of psychotic symptoms on the CAARMS scale
Intensity of psychotic symptoms | 9 months
  Intensity of psychotic symptoms on the CAARMS scale
Distress related to psychotic symptoms | 3 months
  Distress related to psychotic symptoms on the CAARMS scale
Distress related to psychotic symptoms | 4 months
  Distress related to psychotic symptoms on the CAARMS scale
Distress related to psychotic symptoms | 6 months
  Distress related to psychotic symptoms on the CAARMS scale
Distress related to psychotic symptoms | 9 months
  Distress related to psychotic symptoms on the CAARMS scale
Number of patients making a transition to psychosis | 3 months
  Number of patients making a transition to psychosis
Number of patients making a transition to psychosis | 4 months
  Number of patients making a transition to psychosis
Number of patients making a transition to psychosis | 6 months
  Number of patients making a transition to psychosis
Number of patients making a transition to psychosis | 9 months
  Number of patients making a transition to psychosis
Cognitive functions | 3 months
  Cognitive functions measured by the Attentional Performance Tests (APT)
Cognitive functions | 4 months
  Cognitive functions measured by the Attentional Performance Tests (APT)
Cognitive functions | 6 months
  Cognitive functions measured by the Attentional Performance Tests (APT)
Cognitive functions | 9 months
  Cognitive functions measured by the Attentional Performance Tests (APT)
Cognitive functions | 3 months
  Cognitive functions measured by the California Verbal Learning Test (CVLT)
Cognitive functions | 4 months
  Cognitive functions measured by the California Verbal Learning Test (CVLT)
Cognitive functions | 6 months
  Cognitive functions measured by the California Verbal Learning Test (CVLT)
Cognitive functions | 9 months
  Cognitive functions measured by the California Verbal Learning Test (CVLT)
Anxiety | 3 months
  Anxiety measured by the State Trait Anxiety Inventory (STAI)
Anxiety | 4 months
  Anxiety measured by the State Trait Anxiety Inventory (STAI)
Anxiety | 6 months
  Anxiety measured by the State Trait Anxiety Inventory (STAI)
Anxiety | 9 months
  Anxiety measured by the State Trait Anxiety Inventory (STAI)
Functioning | 3 months
  Functioning measured by the Personal and Social Performance Scale (PSP)
Functioning | 4 months
  Functioning measured by the Personal and Social Performance Scale (PSP)
Functioning | 6 months
  Functioning measured by the Personal and Social Performance Scale (PSP)
Functioning | 9 months
  Functioning measured by the Personal and Social Performance Scale (PSP)
Health-related quality of life (HRQoL) | 3 months
  Health-related quality of life (HRQoL) via the SF-12 (12-Item Short Form Health Survey) questionnaire
Health-related quality of life (HRQoL) | 4 months
  Health-related quality of life (HRQoL) via the SF-12 (12-Item Short Form Health Survey) questionnaire
Health-related quality of life (HRQoL) | 6 months
  Health-related quality of life (HRQoL) via the SF-12 (12-Item Short Form Health Survey) questionnaire
Health-related quality of life (HRQoL) | 9 months
  Health-related quality of life (HRQoL) via the SF-12 (12-Item Short Form Health Survey) questionnaire
Health-related quality of life (HRQoL) | 3 months
  Health-related quality of life (HRQoL) via MARS (medication adherence) questionnaire.
Health-related quality of life (HRQoL) | 4 months
  Health-related quality of life (HRQoL) via MARS (medication adherence) questionnaire.
Health-related quality of life (HRQoL) | 6 months
  Health-related quality of life (HRQoL) via MARS (medication adherence) questionnaire.
Health-related quality of life (HRQoL) | 9 months
  Health-related quality of life (HRQoL) via MARS (medication adherence) questionnaire.
Depressive symptoms | 3 months
  Depressive symptoms measured by the Beck Depression Inventory (BDI)
Depressive symptoms | 4 months
  Depressive symptoms measured by the Beck Depression Inventory (BDI)
Depressive symptoms | 6 months
  Depressive symptoms measured by the Beck Depression Inventory (BDI)
Depressive symptoms | 9 months
  Depressive symptoms measured by the Beck Depression Inventory (BDI)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Laprevote, PU.PH, Principal Investigator — Centre Psychothérapique de Nancy
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire (CHU) de Brest, Brest
  - Centre Psychothérapique de Nancy, Laxou

IPD SHARING:
Plan to Share IPD: No